CLINICAL TRIAL: NCT05510973
Title: Evaluation of Advanced HIV Disease Differentiated Care Model in Malawi: A Mixed Methods Non-randomized Cluster Study
Brief Title: Evaluation of Advanced HIV Disease Differentiated Care Model in Malawi
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Elizabeth Glaser Pediatric AIDS Foundation (Other)
Collaborators: Bill and Melinda Gates Foundation (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: EG0264
Record Dates: First submitted 2022-08-15; First posted 2022-08-22 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Opportunistic Infections, HIV-Related; Cryptococcal Infections; AIDS With Tuberculosis; AIDS-related Kaposi Sarcoma; AIDS and Infections
MeSH Terms: conditions — AIDS-Related Opportunistic Infections; AIDS-related Kaposi sarcoma; Acquired Immunodeficiency Syndrome; Infections

STUDY DESIGN:
Intervention Model Description: Non-randomized controlled clustered study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): standard of care
- Intervention (Experimental): Enhanced package of AHD care
  Interventions: Other: Enhanced package for AHD care

INTERVENTIONS:
Other: Enhanced package for AHD care — The enhanced package of AHD care includes CD4 and tuberculosis lipoarabinomannan (TB-LAM) tests and the initiation of patients on TB prophylaxis [TPT and CPT], offered through a hub-and-spoke facility system, with continuous quality improvement (QI)
  Arms: Intervention

SUMMARY:
This study will evaluate the implementation of an enhanced package of care, CD4 and tuberculosis lipoarabinomannan (TB-LAM) tests and the initiation of patients on TB prophylaxis [TPT and CPT], on retention in care and viral suppression ((<50 copies/ml) at 6 and 12 months after AHD care and treatment enrollment. The study will also assess the change in AHD screening, management and service uptake indicators among PLHIV clients before and after implementation of the QI collaborative implementation (QICI) project, evaluate the acceptability and feasibility of the AHD package of care among patients and HCWs providing related health services, and conduct a cost analysis of implementing the enhanced AHD package of care in a hub-and-spoke implementation of care model.

DETAILED DESCRIPTION:
Background Despite significant advances in the diagnosis of human immunodeficiency virus (HIV) and expanded access to anti-retroviral therapy (ART), recent data suggest that a third of people living with HIV/AIDS (PLHIV) starting ART do so with advanced HIV disease (AHD), and an increasing number of patients require advanced HIV disease care following a period of disengagement. Despite considerable effort to implement the AHD model in Malawi and bring it to scale, several challenges regarding AHD implementation and outcomes still exist.

Description of Study Intervention:

To optimize the package of care offered to HIV-infected clients with advanced HIV disease in Malawi, a hub-and-spoke model will be designed and implemented to bring AHD services geographically closer to patients. An enhanced package of AHD interventions such as decentralized cluster of differentiation 4 (CD4) tests, Tuberculosis lipoarabinomannan (TB-LAM) and initiation of patients on prophylaxis [TPT and CPT] will be implemented [system strengthening through quality improvement (QI)]. A client and systems focus will identify challenges experienced by providers and clients while at the same time describing the contextual factors that affect the delivery of AHD services. These lessons learnt will be used to optimize client flow, enhance sample transportation regulation and increase client engagement.

Evaluation Description The evaluation will be a mixed method design study: (1) the quantitative component which will be a non-randomized cluster design based on control of intervention vs control sites for outcomes evaluation (2) the qualitative component that will aim at evaluating acceptability and feasibility of the strengthened AHD service provision (3) cost evaluation that will use quantitative methods.

Specific Objectives

1. To determine the effect of implementation of enhanced AHD package of care in intervention sites versus control sites on the proportion of PLHIV with AHD who are alive and retained in care at 6 and 12 months after diagnosis of AHD and enrolment into AHD care.
2. To determine the effect of implementation of enhanced AHD package of care in intervention sites versus control sites on the proportion of PLHIV with AHD, who achieve viral suppression (<50 copies/ml) at 6 and 12 months after AHD care and treatment enrollment
3. To estimate the change in AHD screening, management and service uptake indicators among PLHIV clients before and after implementation of the QI collaborative implementation (QICI) project
4. To evaluate the acceptability and feasibility of the AHD package of care among patients utilizing AHD services and HCWs providing related health services
5. To conduct a cost analysis of implementing the hub and spoke enhanced AHD package of care to improve AHD differentiated care in selected sites in Malawi.

Endpoints

1. Proportion of PLHIV with advanced disease who will be alive and retained in care at 6 and 12 months after antiretroviral therapy (ART) initiation and after diagnosis of AHD.
2. Proportion of PLHIV with AHD enrolled in care and treatment who are virally suppressed at 6 and 12 months.

Study Population:

The study population for quantitative study component will include children, adolescents and adults of all ages in all the intervention and control sites identified for the project evaluation who are diagnosed with AHD. The study population for the qualitative component will include PLHIV, HCWs and lay cadre supporting the health facility 18 years of age and above available and willing to participate.

Description of Sites/Facilities Enrolling Participants:

The project will be implemented in twenty-two intervention sites in Malawi three selected districts and thirteen control sites in other districts where the intervention is not implemented.

Study duration: The study will take a period of 18 months, including 4 to 6 months enrolment and up to 12 months follow-up.

ELIGIBILITY:
Inclusion Criteria:

HIV-infected clients (all ages) meeting the WHO definition for AHD:

* CD4 count of <200c/mm3
* or WHO clinical stage 3 or 4
* or children under the age of 5 on treatment for less than 12 months or unstable on treatment after 12 months

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 700 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2023-03-31 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of AHD patients alive and retained in care | 6 and 12 months after initiation on ART after AHD diagnosis
  Number of AHD patients alive and retained in care divided by the number of AHD patients initiated on antiretroviral therapy (ART) after diagnosis of AHD
Proportion of AHD patients in care and treatment virally suppressed | 6 and 12 months after initiation of ART after AHD diagnosis
  Number of AHD patients in care and treatment virally suppressed (<50 cells/ml) divided by the number of AHD patients in care and treatment

SECONDARY OUTCOMES:
Cost analysis of implementing the hub and spoke enhanced AHD package of care | 12 months after intervention implementation
  Estimation of total costs, costs per patients with the intervention, and cost drivers

CONTACTS AND LOCATIONS:
Overall Officials: Thulani Maphosa, PhD, Principal Investigator — Elizabeth Glaser Pediatric AIDS Foundation; Appolinaire Tiam, MBChB, MMed, PhD, Principal Investigator — Elizabeth Glaser Pediatric AIDS Foundation; Rose Nyirenda, MPH, PhD, Principal Investigator — Ministry of Health, Malawi
Locations (13):
- Malawi (13):
  - Mlambe Mission Hospital, Mlambe, Blantyre
  - Lobi rural hospital, Lobi, Dedza
  - Mua Mission Hospital, Mtakataka, Dedza
  - Kapiri Mission Hospital, Kapiri, McHinji
  - Domasi Rural Hospital, Domasi, Zomba
  - Chiradzulu District Hospital, Chiradzulu
  - Dedza district hospital, Dedza
  - Mchinji District Hopsital, Mchinji
  - St Michael's Guilleme Community Hospital, Mchinji
  - Ntcheu District Hospital, Ntcheu
  - Sister Theresa Community Hospital, Ntcheu
  - Malamulo Mission Hospital, Thyolo
  - Saint Luke's Mission Hospital, Zomba

REFERENCES:
- [Derived] Katirayi L, Maphosa T, Chilikutali L, Chamanga RK, Petersson J, Khatib S, Munthali B, Nyirenda R, Matiya E, Nyirenda L, Tiam A, Denoeud-Ndam L. Understanding gender differences of people with HIV newly diagnosed or returning to care with advanced HIV disease in Malawi: a qualitative study. BMC Public Health. 2023 Dec 1;23(1):2382. doi: 10.1186/s12889-023-17384-y. PMID 38041058